CLINICAL TRIAL: NCT00001846
Title: Collection and Distribution of Blood Components From Healthy Donors for In Vitro Research Use
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 990168; 99-CC-0168
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-28

CONDITIONS: Blood Donors; Research Subjects; Apheresis
Keywords: Volunteer Donor; Research Samples; Leukapheresis; Plateletpheresis; Plasmapheresis; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- research donors: healthy volunteers (age 18 years or greater) who donate blood for in vitro research purposes

SUMMARY:
This protocol is designed to provide a mechanism for the Department of Transfusion Medicine, Clinical Center to collect and process blood components from paid, healthy volunteer donors for distribution to NIH intramural investigators and FDA researchers for in vitro laboratory use. Donors meeting research donor eligibility criteria will be recruited to donate blood and blood components by standard phlebotomy and apheresis techniques. The investigational nature of the studies in which their blood will be used, and the risks and discomforts of the donation process will be carefully explained to the donors, and a signed informed consent document will be obtained. Donors will be compensated according to an established schedule based on the duration and discomfort of the donation. NIH and FDA investigators requesting blood components for research use will be required to submit an electronic (Web-based) memo of request, briefly describing the nature of the research, and providing assurance that samples provided through this protocol will be used solely for in vitro and not for in vivo research. This protocol also provides a detailed schema for careful and frequent laboratory safety monitoring of repeat research apheresis donors.

Blood components for research use will be distributed with a unique product number, and the DTM principal and associate investigators will serve as the custodians of the code that links the product with a donor s identity. The nature of the in vitro studies in which the blood and components collected in this study will be used is not the subject of this protocol, and is not possible to describe, since it involves basic investigative efforts in greater than 170 different NIH and FDA laboratories. The intent of this protocol is not to approve the research itself, but to provide adequate and complete informed consent for the donor, and to assure that the education, counseling, and protection of the study subjects (research blood donors) is performed in accordance with IRB, OHSR, OPRR and other applicable Federal regulatory standards

DETAILED DESCRIPTION:
This protocol is designed to provide a mechanism for the Department of Transfusion Medicine (DTM), Clinical Center (CC) to collect and process blood components from paid, healthy volunteer donors for distribution to NIH intramural Investigators and FDA researchers for in vitro laboratory use. Donors meeting research donor eligibility criteria will be recruited to donate blood and blood components by standard phlebotomy and apheresis techniques. The investigational nature of the studies in which their blood will be used, and the risks and discomforts of the donation process, will be carefully explained to the donors, and a signed informed consent document will be obtained. Donors will be compensated according to an established schedule, based on the duration and discomfort of their donation. NIH and FDA Investigators requesting blood components for research use will be required to submit an electronic (web-based) memo of request, briefly describing the nature of the research, and providing assurance that samples provided through this protocol will be used solely for in vitro and not for in vivo research. This protocol also provides a detailed schema for careful and frequent laboratory safety monitoring of repeat research apheresis donors.

Blood components for research use will be distributed with a unique product number, and the DTM Principal and Associate Investigators will serve as the custodians of the code that links the product with the donor s identity. The nature of the in vitro studies in which the blood and components collected on this study will be used is not the subject of this protocol, and is not possible to describe since it involves basic investigative efforts in greater than multiple different NIH and FDA laboratories. The intent of this protocol is not to approve the research itself, but to provide adequate and complete informed consent for the donor, and to assure that the education, counseling, and protection of the study subjects (research blood donors) are performed in accordance with the Institutional Review Board (IRB), the Office of Human Subjects Research Protection (OHSRP), and other applicable Federal regulatory standards.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Donors must meet the eligibility criteria for volunteer blood donation, defined in the Code of Federal Regulations 21 CFR 640, and AABB Standards as modified in the 2007 FDA/CBER Guidance Document: Eligibility Criteria for Donors of Human Cells, Tissues, and Cellular and Tissue-Based Products, with the exception of foreign travel history and other conditions, as noted below:

* Ability of subject to understand, ask questions, and the willingness to provide written informed consent
* Age greater than or equal to 18 years
* Weight greater than 110 pounds
* Female subjects should not be pregnant
* No known heart, lung, kidney disease, or bleeding disorders
* No history of sickle cell disease
* No history of engaging in high-risk activities for exposure to the AIDS virus, as defined in the AABB Donor Education Materials distributed to all donors. Deferral periods for high-risk activities (MSM, IV drug use or receipt of money or drugs in exchange for sex) will not exceed the corresponding deferral period as defined for allogeneic blood donors.
* No history of malaria in the past 12 months
* Donors who have a family history of CJD, donors who have undergone tattooing or body piercing, donors who have received a graft such as bone, skin or dura mater, donors who are taking finasteride or retinoids, and donors who have had sexual contact within the past 12 months with a person who has symptomatic hepatitis C infection or donors who have lived with a person who has hepatitis in the last 12 months, are similarly eligible for research-use only donations on this protocol.
* Donors who have traveled to Europe, Africa, Asia, and areas of South America, who are rendered ineligible for allogeneic donation due to malarial risk, Zika risk and vCJD risk, are eligible for research donations
* Donors with a history of repeat false positive HTLV I/II, who are rendered ineligible for allogeneic donation, are eligible for research donations.
* Donors with a positive antibody to hepatitis B core antigen (anti-HBc) only, without other positive infectious disease markers,are eligible for research donations.
* Donors with HLA antibodies are eligible for research donations
* Donors who have received an experimental drug, agent, or vaccine, and who are referred for a research blood, plasma or leukocyte collection, specifically because they were given this drug, agent, or vaccine, are acceptable only if their research product is collected for use by the PI who administered the experimental drug, agent, or vaccine. Otherwise, they are deferred for one year after receiving an experimental drug, agent, or vaccine.
* Donors who have received a xenotransplant are eligible for research donations.
* Granulocyte donors may not receive dexamethasone if they have poorly controlled hypertension or diabetes, or if they have a history of cataracts. Hetastarch (also known as hydroxyethyl starch or "HES") and dexamethasone may elevate blood pressure and raise blood glucose levels, and repetitive steroid administration may increase the risk of posterior subcapsular cataract formation or progression.
* Granulocyte donors must have an estimated glomerular filtration (eGFR) rate of > 45ml/min/1.73m^2.
* Granulocyte donors may not receive filgrastim if they have a history or symptoms of coronary heart disease.

Investigators are informed that eligibility standards for research donors differ from those for transfusion donors through an electronic "User Agreement" which they electronically sign when they register to receive blood components on this protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer donors
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2001-01-11 (Actual)

PRIMARY OUTCOMES:
Provision of samples to researchers | Quarterly
  Provision of samples to researchers

CONTACTS AND LOCATIONS:
Overall Officials: Kamille A West-Mitchell, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Nishio K, Pasquet L, Camara K, DiSapio J, Hsu KS, Kato S, Bloom A, Richardson SK, Welsh JA, Jiang T, Jones JC, Cardell S, Watarai H, Terabe M, Olkhanud PB, Howell AR, Berzofsky JA. Lysosomal processing of sulfatide analogs alters target NKT cell specificity and immune responses in cancer. J Clin Invest. 2023 Dec 21;134(4):e165281. doi: 10.1172/JCI165281. PMID 38127463
- [Derived] Dahut M, Fousek K, Horn LA, Angstadt S, Qin H, Hamilton DH, Schlom J, Palena C. Fulvestrant increases the susceptibility of enzalutamide-resistant prostate cancer cells to NK-mediated lysis. J Immunother Cancer. 2023 Sep;11(9):e007386. doi: 10.1136/jitc-2023-007386. PMID 37678915
- [Derived] Han K, Singh K, Meadows AM, Sharma R, Hassanzadeh S, Wu J, Goss-Holmes H, Huffstutler RD, Teague HL, Mehta NN, Griffin JL, Tian R, Traba J, Sack MN. Boosting NAD preferentially blunts Th17 inflammation via arginine biosynthesis and redox control in healthy and psoriasis subjects. Cell Rep Med. 2023 Sep 19;4(9):101157. doi: 10.1016/j.xcrm.2023.101157. Epub 2023 Aug 15. PMID 37586364
- [Derived] Cho YE, Lee H, Bae HR, Kim H, Yun S, Vorn R, Cashion A, Rucker MJ, Afzal M, Latour L, Gill J. Circulating immune cell landscape in patients who had mild ischaemic stroke. Stroke Vasc Neurol. 2022 Aug;7(4):319-327. doi: 10.1136/svn-2021-001224. Epub 2022 Mar 9. PMID 35264400
- [Derived] Horn LA, Chariou PL, Gameiro SR, Qin H, Iida M, Fousek K, Meyer TJ, Cam M, Flies D, Langermann S, Schlom J, Palena C. Remodeling the tumor microenvironment via blockade of LAIR-1 and TGF-beta signaling enables PD-L1-mediated tumor eradication. J Clin Invest. 2022 Apr 15;132(8):e155148. doi: 10.1172/JCI155148. PMID 35230974
- [Derived] Wu J, Singh K, Lin A, Meadows AM, Wu K, Shing V, Bley M, Hassanzadeh S, Huffstutler RD, Schmidt MS, Blanco LP, Tian R, Brenner C, Pirooznia M, Kaplan MJ, Sack MN. Boosting NAD+ blunts TLR4-induced type I IFN in control and systemic lupus erythematosus monocytes. J Clin Invest. 2022 Mar 1;132(5):e139828. doi: 10.1172/JCI139828. PMID 35025762
- [Derived] Han K, Singh K, Rodman MJ, Hassanzadeh S, Wu K, Nguyen A, Huffstutler RD, Seifuddin F, Dagur PK, Saxena A, McCoy JP, Chen J, Biancotto A, Stagliano KER, Teague HL, Mehta NN, Pirooznia M, Sack MN. Fasting-induced FOXO4 blunts human CD4+ T helper cell responsiveness. Nat Metab. 2021 Mar;3(3):318-326. doi: 10.1038/s42255-021-00356-0. Epub 2021 Mar 15. PMID 33723462
- [Derived] Donahue RN, Lepone LM, Grenga I, Jochems C, Fantini M, Madan RA, Heery CR, Gulley JL, Schlom J. Analyses of the peripheral immunome following multiple administrations of avelumab, a human IgG1 anti-PD-L1 monoclonal antibody. J Immunother Cancer. 2017 Feb 21;5:20. doi: 10.1186/s40425-017-0220-y. eCollection 2017. PMID 28239472
- [Derived] Maynard DM, Heijnen HF, Gahl WA, Gunay-Aygun M. The alpha-granule proteome: novel proteins in normal and ghost granules in gray platelet syndrome. J Thromb Haemost. 2010 Aug;8(8):1786-96. doi: 10.1111/j.1538-7836.2010.03932.x. Epub 2010 May 27. PMID 20524979
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1999-CC-0168.html